CLINICAL TRIAL: NCT00469027
Title: Phase I Trial to Establish Safety of Autologous Progenitor Cell-based Gene Therapy Delivery of heNOS in Patients With Severe Pulmonary Arterial Hypertension(PAH)Refractory to Conventional Treatment
Brief Title: Pulmonary Hypertension: Assessment of Cell Therapy
Acronym: PHACeT
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Northern Therapeutics (Industry)
Collaborators: Unity Health Toronto (Other); Sir Mortimer B. Davis - Jewish General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: CT-PAH 001
Record Dates: First submitted 2007-05-02; First posted 2007-05-04 (Estimated); Last update posted 2016-10-17 (Estimated); Status verified 2016-10

CONDITIONS: Hypertension, Pulmonary
Keywords: Pulmonary Arterial Hypertension (PAH)
MeSH Terms: conditions — Hypertension, Pulmonary; Pulmonary Arterial Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- eNOS transfected EPCs (Experimental): eNOS transfected EPCs will be delivered by injection via a PA line, incremental doses over three days
  Interventions: Biological: eNOS transfected EPCs will be delivered via a PA line

INTERVENTIONS:
Biological: eNOS transfected EPCs will be delivered via a PA line — incremental dosing over 3 days
  Other Names: eNOS transfect EPCs

SUMMARY:
The primary objective is to establish the safety of autologous progenitor cell-based gene therapy of heNOS in patients with severe Pulmonary Arterial Hypertension(PAH) refractory to conventional treatment.

DETAILED DESCRIPTION:
This is a two centre, phase I clinical trial. A total of 18 patients will be studied using an open-label, dose escaling protocol; three patients will be entered into each of the five dosing panels. An additional three patients will be entered into the final dose panel to establish safety at the maximum tolerated dose.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of idiopathic Pulmonary Arterial Hypertension
* Familial PAH or anorexigen induced PAH
* Specified 6-minute walk distance

Exclusion Criteria:

* Intra or extra cardiac communication between the right and left sided circulations
* Hemodynamic instability
* Left ventricular ejection fraction < 40%
* Thromboembolic event or recent hospitalization for worsening right sided heart failure in past 3 months
* CVP>20mmHg at time of research heart catheterization
* Pregnancy
* Concurrent hepatitis or HIV

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2006-05; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
The primary endpoints will be related to the tolerability and safety of injection of genetically engineered progenitor cells in patients with severe PAH. | 5 years

SECONDARY OUTCOMES:
Potential efficacy of this approach will be assessed by changes in hemodynamic pressures, patient perceived quality of life and exercise capacity | 3 month post cell delivery

CONTACTS AND LOCATIONS:
Overall Officials: John Granton, MD, Principal Investigator — St. Michael's Hospital and University Health Network; David Langleben, MD, Principal Investigator — Sir Mortimer B. Davis - Jewish General Hospital
Locations (2):
- Canada (2):
  - St. Michael's Hospital, Toronto, Ontario
  - Sir Mortimer B. Davis - Jewish General Hospital, Montreal, Quebec

REFERENCES:
- [Derived] Granton J, Langleben D, Kutryk MB, Camack N, Galipeau J, Courtman DW, Stewart DJ. Endothelial NO-Synthase Gene-Enhanced Progenitor Cell Therapy for Pulmonary Arterial Hypertension: The PHACeT Trial. Circ Res. 2015 Sep 11;117(7):645-54. doi: 10.1161/CIRCRESAHA.114.305951. Epub 2015 Jul 20. PMID 26195220
- [Derived] O'Connell C, O'Callaghan DS, Humbert M. Novel medical therapies for pulmonary arterial hypertension. Clin Chest Med. 2013 Dec;34(4):867-80. doi: 10.1016/j.ccm.2013.08.002. PMID 24267310